CLINICAL TRIAL: NCT02084732
Title: Safety and Efficacy of Sorafenib in Patients With Advanced Thyroid Cancer: a Phase II Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 410-30610-258
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Thyroid Cancer
Keywords: Sorafenib, thyroid neoplasms, salicylic acid
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): drug
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — drug
  Other Names: nexavar

SUMMARY:
Differentiated thyroid cancer includes papillary, follicular, Hurthle cell, and C-cell/medullary carcinoma. Even though incidence is relatively low (1% of all neoplasms), a rise in this disease has been recorded in the country (The Atlas of Cancer Mortality in Colombia, 2010).

Although this disease has a low rate of attributable mortality, the costs arising from treatment, monitoring, and disabilities among affected patients and their families are high for the health system.

The therapeutic approach to differentiated thyroid cancer once it starts progressing is limited; there are no truly favorable treatment options for patients with advanced thyroid cancer: available options include surgery, radiotherapy, and radioactive iodine therapy.

Molecular biology now allows the identification of the effects of mutations and alterations in the proteins that participate in cell signaling which account for dedifferentiation, invasiveness, and the progression of neoplastic cells.

VEGFR (vascular endothelial growth factor receptor) is one of the main molecules to be addressed by targeted molecular therapy. Its increased expression in differentiated thyroid cancer has been demonstrated and has been associated with increased growth, invasiveness, and shorter recurrence-free survival.

Different agents are effective against this tyrosine kinase receptor; nevertheless, taking into account that it is not solely responsible for tumor progression, according to clinical study results, it is more reasonable to use non-selective tyrosine kinase inhibitors such as sorafenib and motesanib. These inhibitors have already been tested in phase II studies.

Results from recent phase II research studies using these emerging treatment options have shown important effects in the therapeutic approach to other solid neoplasms.

Information about the safety of this type of treatment is limited; a need for information regarding the use of new therapeutic approaches in Colombia is one of the contributions that the National Institute of Cancer can make to the country through this study.

DETAILED DESCRIPTION:
Objective:

Determine the clinical efficacy and safety profile of sorafenib in the treatment of patients with advanced thyroid cancer (metastatic or recurrent) in a 24 months follow up period.

Analysis plan The analysis plan includes the description of clinical and epidemiological characteristics of recruited patients at the end of the first year and the before and after comparison from clinical response according to RECIST criteria. At the end of the first and second follow-up years, analyses will be performed. In each of these, the response of patients by outcomes of interest measured at specific monitoring times will be evaluated.

Parametric and non-parametric descriptive statistics will be used as necessary; the comparison of some variables between baseline measurements and follow-up predetermined cut-offs will be performed while taking into account the lack of independence between observations. Analysis of qualitative variables will be performed using McNemar's Test and the analysis of quantitative variables using the Paired Student's t-Test or Wilcoxon Test depending on the normality of the distribution

Descriptive statistics will be used for time until events, survival curve and progression-free time median will be stated. Correlation studies between some indicators, clinical variables, and observed outcomes using parametric and non-parametric coefficients will be performed. Interobserver agreement will be evaluated for the reading of diagnostic images using a Kappa coefficient.

ELIGIBILITY:
* Older than 18 years.
* Confirmed histological diagnosis of differentiated thyroid cancer, whether metastatic or unresectable, for whom conventional curative or palliative therapeutic options do not exist or are not effective. It includes patients with lesions visible in images, that have no uptake at therapeutic doses of iodine, or patients with iodine avid lesions, that keep progressing after therapeutic doses (greater than 100 mCi). Also comprises patients with persistent local disease progression not amenable to surgical management or radiation therapy management.
* The time that has passed since the last treatment until inclusion must of at least six (6) months.
* There must be at least 1 lesion that can be adequately measured according to the RECIST (v.1.1) criteria [See Appendix 1].
* Neck or lung lesions, surgery declared unresectable.
* Patients must have a ECOG score less than 2 and life expectancy greater than 3 months.
* Adequate bone marrow, liver and renal functions defined by the following laboratory parameters, taken no more than 7 days after consent signing: white blood cell count, > 3,000/uL; absolute neutrophil count, > 1,500/mm3; platelets, > 100,000/mm3; hemoglobin, 9 g/dl; serum creatinine, < 1.5 times the upper limit of normal (ULN) or creatinine clearance in urine for 24 hours > 75 cc/min; total serum bilirubin, < 1.5 times the ULN; glutamic oxaloacetic transaminase (SGOT), < 1.5 times the ULN; serium alkaline phosphatase, < 1.5 times the ULN; prothrombin time (PT-INR) and partial thromboplastin time (PTT), < 1.5 times the ULN.
* The patient must be physically, intellectually, and emotionally able to take the oral medicine.
* Patient must not be a candidate for surgery or radiotherapy with curative intent
* Women of childbearing potential should have a negative serum pregnancy test performed within 7 days prior to start of treatment. Post-menopausal women (at least one year with no menstruation) and surgically sterilized women do not require pregnancy tests.
* Women and also men of childbearing potential should agree to use adequate contraceptive methods
* Significant medical conditions including an uncontrolled hypertension (systolic blood blood pressure >150 mmHg or diastolic blood pressure > 90mmHg)
* Significant Hemorrhage or bleeding events, CTCAE grade 3 or higher, within 12 weeks of randomization. arterial or venous thrombotic or embolic events within the past 6 months (including cerebrovascular accidents and transient ischemic attacks, deep vein thrombosis, pulmonary embolism and arterial thrombosis).
* Recent major surgery or open biopsy procedure (within 4 weeks of study entry)
* Bone lesions will be excluded, by its susceptibility to radiotherapy and bisphosphonates management.
* Wounds, ulcers or bone fractures that are non healing
* Pregnancy or lactation.
* A personal history of a second neoplasm with the exception of squamous-cell or basal-cell skin cancer that is suitably treated, in situ cervical cancer, or any other previously treated cancer when one has stayed free of disease for 5 years or more.
* Prior use (4 weeks before admittance to the study) of chemotherapy or cancer immunotherapy.
* Prior use of of tyrosine kinase inhibitors or other targets agents, or monoclonal antibodies that target VEGF or VEGF receptors.
* Known or suspected allergy or hypersensitivity to sorafenib
* Having received radiotherapy in the 4 weeks preceding admittance to the study.
* Any condition according to the judgment of the treating physician that could jeopardize the patient's safety or compliance to the study.
* All patients that are admitted to the study must voluntarily consent to their participation and the same must be recorded in a written informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Describe the clinical activity and safety profile of sorafenib in the treatment of patients with advanced thyroid cancer (metastatic or recurrent) among a selected group of patients refractory to or ineligible to radioactive iodine (RAI) therapy | 3 years

SECONDARY OUTCOMES:
Summarize the progression-free survival (PFS) of patients with advanced thyroid cancer (metastatic or recurrent) treated with sorafenib | two years
Describe the occurrence and type of adverse events associated with sorafenib use in advanced thyroid cancer (metastatic or recurrent) patients included | two years

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Fierro, Md, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerología, Bogotá, Cundinamarca, Colombia